CLINICAL TRIAL: NCT00266279
Title: Phase II Study of Oxaliplatin and Capecitabine in Advanced Head and Neck Malignancies
Brief Title: Phase II (Treatment) Study of Oxaliplatin and Capecitabine in Advanced Head and Neck Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 153.05
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Head or Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with Study Drugs (Experimental): Treatment with combination of oxaliplatin and capecitabine using study dose and schedule.
  Interventions: Drug: Oxaliplatin, Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin, Capecitabine — Agent, DOSE AND SCHEDULE (28-days cycle):
  Oxaliplatin 85 mg/m2 IV on days 1 and 15 Capecitabine 1500 mg PO BID on days 1-7 and 15-21

SUMMARY:
This phase II study will test the response rate of combined oxaliplatin and capecitabine treatment when administered at a given dose and schedule, in patients with Head and Neck cancer for which there is no curative treatment.

DETAILED DESCRIPTION:
The optimal dose and schedule for the combined treatment with oxaliplatin and capecitabine have not been defined. The aim of this Phase II study is to determine the response rate of combined oxaliplatin and capecitabine treatment at a given dose and schedule in patients with Head and Neck cancer for which there is no curative treatment.

The study also aims to determine the qualitative and quantitative toxicity and reversibility of toxicity of the above combination and to evaluate any changes in performance status, quality of life, overall survival and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell cancer of Head and Neck
* Patients must have metastatic or locally recurrent disease
* Patients must have disease not curable by surgery as estimated by one of the protocol investigators, and should not be eligible for reradiation protocol or have failed reradiation protocol.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan
* Age >18 years of age
* Life expectancy of greater than 12 weeks
* ECOG performance status 0, 1 or 2 (Karnofsky >50%; see Appendix B)
* Patients must have adequate bone marrow function as defined below:

  * absolute neutrophil count > 1,500
  * platelets > 100,000
  * hemoglobin > 8 g/dl
* Patients must have adequate renal function as defined by a creatinine clearance >30 mL/min (measured or estimated by the Cockroft and Gault equation)

  * Cockroft and Gault equation:
  * Creatinine clearance for males =(140-age[yrs])(body wt[kg])/72(serum creatinine[mg/dL])
  * Creatinine clearance for females = 0.85 x male value
* Patients must have adequate liver function as defined below:

  * total bilirubin 1.5x upper limit of normal
  * albumin > 2.5 g/dl
  * AST(SGOT) and ALT(SGPT) and Alkaline Phosphatase must be < 5 times upper limit of normal
* Patients could have received 1 or 2 previous chemotherapy regimens prior to entering the study. Patients must have recovered from acute toxicities from chemotherapy or radiotherapy administered prior to entering this study. Alopecia may not be resolved and peripheral neuropathy (grade 1) may be present.
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil or oxaliplatin
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to first treatment in this study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients receiving any other investigational agent(s)
* Patients with symptomatic brain metastases or actively receiving any therapy for brain metastasis (because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events)
* Active second malignancy in the last 5 years except for non-melanoma skin cancer or carcinoma-in-situ
* Clinically significant cardiac disease (e.g. congestive heart failure, New York Heart Association Class II or greater, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months.
* If patient is unable to swallow, xeloda may be crushed per hospital policy/procedure. See attached Appendix G.
* Patients who have had an organ allograft.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy
* Known Hepatitis B , Hepatitis C, HIV

Inclusion of Minorities:

Members of all ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damian Laber, M.D., Principal Investigator — University of Louisville, James Graham Brown Cancer Center
Locations (1):
- University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Result] Rabinowits G, Bhupalam L, Miller DM, Kloecker GH, Laber DA. Fixed-dose every-other-week capecitabine and oxaliplatin for refractory squamous cell carcinoma of the head and neck. Am J Med Sci. 2010 Feb;339(2):148-51. doi: 10.1097/MAJ.0b013e3181c4bd91. PMID 20087165
- See also: James Graham Brown Cancer Center website — http://browncancercenter.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With Study Drugs: Treatment with combination of oxaliplatin and capecitabine using study dose and schedule.
  Oxaliplatin, Capecitabine : Agent, DOSE AND SCHEDULE (28-days cycle):
  Oxaliplatin 85 mg/m2 IV on days 1 and 15 Capecitabine 1500 mg PO BID on days 1-7 and 15-21
Period: Overall Study
Arm/Group | Treatment With Study Drugs
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Study Drugs
Number analyzed (Participants) | 15
Age, Customized [Number; unit: Participants]
  >=18 years | 15
Sex/Gender, Customized [Number; unit: Participants]
  Male | 10
  Femal | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Among the 15 patients treated, 2 (13%) achieved partial response (PR), and 5 (33%) achieved stable disease (SD), for a Overall Response Rate (ORR) of 46% measured by RECIST criteria.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  Overall Response Rate (ORR)=PR+CR.
Time Frame: Every two 28 day treatment cycles until subject no longer on treatment due to disease progression
Measure: Number; unit: Participants
Arm/Group | Treatment With Study Drugs
Number analyzed (Participants) | 15
Participants
  Partial Response | 2
  Stable Disease | 5

2. Secondary Outcome: Qualitative and Quantitative Toxicity
Description: Number of patients that developed common side effect of diarrhea.
Time Frame: At study enrollment, Every two 28 day treatment cycles, and at end of treatment due to disease progression
Measure: Number; unit: participants
Groups:
- Treatment With Study Drugs: Treatment with combination of oxaliplatin and capecitabine using study dose and schedule.
  Oxaliplatin, Capecitabine: Agent, DOSE AND SCHEDULE (28-days cycle):
  Oxaliplatin 85 mg/m2 IV on days 1 and 15 Capecitabine 1500 mg PO BID on days 1-7 and 15-21
Arm/Group | Treatment With Study Drugs
Number analyzed (Participants) | 15
participants | 2

ADVERSE EVENTS:
Arm/Group | Treatment With Study Drugs
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Study Drugs (N=15)
Pneumonia (Infections and infestations) | 2 (2) — Two patients were hospitalized because of pneumonia.
Dehydration (General disorders) | 1 (1) — 1 subjects was hospitalized for dehydration.
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) — 1 Subject experienced gastrointestinal bleeding.

LIMITATIONS AND CAVEATS:
Results data not available, PI not longer at institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No